CLINICAL TRIAL: NCT00931567
Title: Evaluation of the Efficiency of Autologous Platelet Gel (Platelet Rich Fibrin) Obtained From Own Patients' Blood Versus Vaselitulle in Dupuytren's Disease Postoperative Wound Healing
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: University Hospital, Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-APR-07
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Dupuytren's Contracture
MeSH Terms: conditions — Dupuytren Contracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vaselitulle (Active Comparator): after surgery, the loss of substance is treated using vaseline dressing
  Interventions: Device: Vaselitulle
- Autologous platelets gel (Experimental): after surgery, the loss of substance is treated with Autologous platelets gel
  Interventions: Biological: Autologous platelets gel

INTERVENTIONS:
Biological: Autologous platelets gel — Application of autologous platelets gel (Platelet Rich Fibrin) after the " open palm " surgical treatment of Dupuytren's disease.
  Arms: Autologous platelets gel
Device: Vaselitulle — application of standardized wound dressing after the " open palm " surgical treatment of Dupuytren's disease.
  Arms: Vaselitulle

SUMMARY:
This study is a clinical, multicentric, randomised open trial. The objective is to evaluate the efficiency, in terms of wound healing speed, of peroperative application of autologous platelets gel versus standardized wound dressing. The wound Healing model used in this study is the " open palm " surgical treatment of Dupuytren's disease.

Dupuytren's disease is a fibroproliferative disease of the palmar and digital fascia of the hand that may lead to a fixed flexion contracture of the fingers.

The main indication for surgery is the loss of finger extension. In some cases of palmar Dupuytren's disease the surgical removal of diseased tissues may lead to a cutaneous loss of substance (" open palm technique "). This loss of substance is treated using vaseline dressing and the wound healing is obtained in 4 weeks.

Autologous platelets gel (Platelet Rich Fibrin) is obtained from the patient's own blood. Some recent studies have shown that it speeds up the wound healing and enhances the quality of the scar.

PRF belongs to a new generation of autologous platelet gel that are easily obtained after centrifugation of patient's own blood.

The Platelet Rich Fibrin (PRF) contains many wound healing factors : Three pro inflammatory cytokines ( IL1,IL6, TNF-alpha) , one anti-inflammatory cytokine (IL4) and a growth factor (VEGF).

The study will be running on 60 days, starting from the operation day. The wound healing evaluation will be achieved at day1, day2, day7, day14, day 21 day 28 and day 60.

The inclusion criteria are : age over 18, Dupuytren's disease with an indication of surgical treatment using the open palm technique, patients having signed the agreement form.

80 patients will be included in the study and divided into 2 groups . The first group of patients will receive PRF and the other group will receive vaseline dressings.

The speed and the quality of wound healing will be compared.We will also compare the number of patients with a complete wound healing at day 21 . Moreover,we will evaluate the pain during the dressings' change and the bleeding of the palmar wound.

For the wound healing speed , a difference of 7 days between the two groups will be considered as statistically significant.

Statistical analysis will be achieved using Chi2 test and Logrank test.

DETAILED DESCRIPTION:
Main evaluation criteria :

Time duration between the operation and the complete wound healing. The wound healing is considered complete when the skin is closed and when the patient do not need to have dressings. A picture of the wound at the end of the wound healing process is taken for each patient.

Secondary criteria of evaluation :

At day 1, day7, day 14, day 21 and day 28 two data will be collected :

* The pain during the dressings' change using a visual scale going from 0 (no pain) to 10 (very painful).
* The bleeding (and "exudate") of the wound which can be absent, low, moderate or abundant.

The investigators will collect all the side effects described by the patients for each wound healing technique.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Patient with Dupuytren's disease with an indication of surgical treatment using the open palm technique.
* Agreement form signed
* patient affiliated to the national health system.

Exclusion Criteria:

* Patients allergic to one of the components of the dressings used in this study.
* Patients with insulin-requiring diabetes
* Patients sustaining anti-cancer treatment.
* Pregnant women.
* Patients included in another study.
* Patients who cannot come to the follow up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-08; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Time duration between the operation and the complete wound healing. | 18 months

SECONDARY OUTCOMES:
-The pain during the dressings' change using a visual scale going from 0 to 10. -The bleeding of the wound. | 18 months

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Hôpital de la Timone, Marseille, Cedex 05
  - Centre Hospitalier Universitaire de Nice Hôpital de Cimiez, Nice

REFERENCES:
- [Derived] Chignon-Sicard B, Georgiou CA, Fontas E, David S, Dumas P, Ihrai T, Lebreton E. Efficacy of leukocyte- and platelet-rich fibrin in wound healing: a randomized controlled clinical trial. Plast Reconstr Surg. 2012 Dec;130(6):819e-829e. doi: 10.1097/PRS.0b013e31826d1711. PMID 23190833